CLINICAL TRIAL: NCT06709976
Title: Increasing the Accuracy to Predict Pregnancy Success After Assisted Reproductive Therapy (ART) by Combining the ReceptIVFIty Test with Immunological Parameters
Brief Title: ReceptIVFity & Immunology in ART
Acronym: R-IMinART
Status: Enrolling by invitation | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Sam Schoenmakers, Principal Investigator, Erasmus Medical Center
Other Study IDs: OZBS72.19236
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-09

CONDITIONS: Infertility (IVF Patients); Infertility Assisted Reproductive Technology
Keywords: IVF success prediction; Vaginal microbiome; Menstrual blood immunology; Assisted reproductive technology (ART); Infertility biomarkers
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal microbiome sample Self-collected Menstrual Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Vaginal microbiome swab — All swabs were collected using FLOQSwabs™ (Copan Italia SpA, Brescia, Italy). The patients were instructed to spread the labia with one hand, insert the swab 3-5 cm beyond the vaginal orifice with the other hand, and rotate the swab along the vaginal wall for 10-15 seconds.
Device: Menstrual Blood Collection via Menstrual Cup — Self-collect menstrual blood during 24 hours in 2 blocks of 12 hours

SUMMARY:
The goal of this clinical non-invasive observational pilot study is to improve the prediction of pregnancy success after In Vitro Fertilisation (IVF)/IVF -Intracytoplasmic Sperm Injection (ICSI) treatment by examining the vaginal microbiome and the immunological profile of menstrual blood in women (18-42) years old) undergoing their first IVF/IVF/ICSI treatment.

The main questions it aims to answer are:

What is the ReceptIVFity profile (low, medium, or high) of the vaginal microbiome in these women? How do the endometrial-derived lymphocytes respond to different immune stimuli and microbiota? Can the endometrial stromal cells decidualize effectively in the presence or absence of specific microbiota?

Participants will:

Self-perform a vaginal swab to determine the ReceptIVFity profile of their vaginal microbiome.

Self-collect menstrual blood during 24 hours in 2 blocks of 12 hours for immunological analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Indication for an IVF or IVF/ICSI procedure.
2. 18 years - 42 years.
3. European origin
4. Willing to provide a vaginal swab with the ReceptIVFity-test.
5. Willing to provide informed consent.

Exclusion Criteria:

1. No transferable embryos after IVF or IVF/ICSI.
2. Emergency IVF for cancer or other reasons.
3. Women with endometriosis pre-treated with an Gn-RH analogue.
4. The use of (hormonal) contraceptives or antibiotics 3 months prior to start IVF or IVF/ICSI.
5. Women unable or unwilling to agree with the procedures.
6. Women unable or unwilling to give written informed consent.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who receive IVF or IVF/ICSI treatment
Study Population: Women aged 18-42 expected to undergo their first IVF/IVF-ICSI cycle within the next two months. The routine IVF/IVF-ICSI procedure will occur irrespective of their participation or the test outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Immune Cell Phenotype and Function in Menstrual Blood Stratified by Vaginal Microbiome in IVF Patients | Baseline and 3 months
  Analysis of monocyte, Natural Killer (NK) cell, T lymphocytes, regulatory T lymphocytes, and T helper cell phenotypes in menstrual blood. Immune responses, including cytokine production and immune marker regulation, will be quantified.
  Unit of Measure: Percentage of cell type, cytokine concentrations in pg/mL.
Genotyping of Maternal KIR and HLA-C | Baseline
  Determination of maternal Killer cell immunoglobulin-like receptor (KIR) and Major Histocompatibility Complex (HLA-C) genotypes.
  Unit of Measure: Genotype classification.
RNA Analysis of Stromal Fibroblast Cells | Baseline
  Analysis of RNA from stromal fibroblast cells to determine expression of tissue adaptation markers (pre-decidualization).
  Gene expression levels (e.g., fold change, normalized counts).

SECONDARY OUTCOMES:
Metabolite Analysis as Immune Signaling Modulators in IVF Patients | Baseline
  Analysis of host- and microbiome-derived metabolites serving as signaling molecules that regulate immune function.
  Unit of Measure: Metabolite concentrations (µmol/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No